CLINICAL TRIAL: NCT04418388
Title: A Single Center, Open-label Clinical Trial to Evaluate Pharmacokinetic Characteristics and Safety of PBK-1801 After Single Oral Administration in Healthy Korean Women Volunteers
Brief Title: Pharmacokinetics and Safety of PBK-1801 After Single Oral Administration in Healthy Korean Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmbio Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PBK_1801_101
Record Dates: First submitted 2020-05-26; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- A (Experimental)
  Interventions: Drug: PBK-1801
- B (Experimental)
  Interventions: Drug: PBK-1801
- C (Experimental)
  Interventions: Drug: PBK-1801

INTERVENTIONS:
Drug: PBK-1801 — Administered orally
  Arms: A
Drug: PBK-1801 — Administered orally
  Arms: B
Drug: PBK-1801 — Administered orally
  Arms: C

SUMMARY:
The primary objective of this study is to assess the pharmacokinetic characteristics after a single dose of oral PBK-1801 in healthy Korean women for preparing the bridging data for Koreans.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 19 and 30 kg/m²
* Subjects are to be in good general health according to medical history, physical examination, electrocardiograph (ECG) recording and clinical laboratory assessments showing no signs clinically significant pathology (A subject with a clinically insignificant abnormality may be included by the discretion of the investigator)
* Subjects are to have given their written informed consent to participate in the study and to abide by study restrictions

Exclusion Criteria:

* History or evidence of clinically significant cardiovascular, renal, hepatic, hematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological, psychiatric or other major disease
* Subjects who have any condition possibly affecting drug absorption (e.g., previous surgery on the gastrointestinal tract other than uncomplicated appendectomy, inflammatory bowel disease).
* History or current alcohol abuse or drug addiction
* Subjects who for any reason, are deemed by the Investigator to be inappropriate for this study

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Cmax | 5 days
AUClast | 5 days
AUCinf | 5 days
Tmax | 5 days
T1/2 | 5 days
CL/F | 5 days
Vd/F | 5 days

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: SeungHwan Lee, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea